CLINICAL TRIAL: NCT03093558
Title: Pilot Atrial Fibrillation Information Technology Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jared W Magnani, MD, MSc, Associate Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO16020290
Record Dates: First submitted 2017-03-02; First posted 2017-03-28 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Atrial Fibrillation
Keywords: adherence; quality of life; health literacy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Receive the ECA/Kardia for 30-day use.
  Interventions: Behavioral: ECA/Kardia
- Usual care arm (No Intervention): Receive a journal for observation of adherence and symptoms.

INTERVENTIONS:
Behavioral: ECA/Kardia — Use of the ECA and Kardia daily for 30 days.
  Arms: Intervention arm

SUMMARY:
AF is associated with significant social and medical costs, including diminished quality of life (QOL) and increased health care utilization (HCU). This pilot study will enroll 200 adults with prevalent, non-valvular AF of ≤3 year's duration at University of Pittsburgh Medical Center (UPMC). The primary objective at present is to obtain extensive feasibility and pilot data in implementing the Embodied Conversational Agent (ECA) in concert with the Kardia (KAC) heart rhythm monitor.

DETAILED DESCRIPTION:
This pilot study is a single-center, two-arm randomized study that by design is unblinded. 200 total participants are planned. Each participant will be randomized in an unblocked manner to receive "usual care" or the ECA/KAC intervention. Participants will have study visits at baseline and time 30 days. Adherence to using the ECA/KAC in combination over 30 days will be quantified. Following participation study participants randomized to the ECA/KAC intervention will undergo an interview to determine their experience with the ECA/KAC. Participants and their physicians will receive a summary of ECA use and symptoms and correlated findings by KAC.

ELIGIBILITY:
Inclusion Criteria:

* CHADS2-VASc score ≥2; English-speaking (at level appropriate to provide informed consent and participate in this research protocol); no plan to relocate from the area within 12 months of enrollment

Exclusion Criteria:

* AF that is due to non-cardiac causes (e.g., sepsis, pneumonia, thyroid disorders, and intoxication); AF within 30 days of any cardiothoracic or thoracic surgery; Inability to complete training session with the smartphone and demonstrate use of the ECA; Inability to answer specific protocol-based questions correctly during consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Daily adherence to the Embodied Conversational Agent and Kardia heart rhythm monitor | 30 days
  Assessment of daily use of the combined ECA and Kardia heart rate/rhythm monitor

SECONDARY OUTCOMES:
Participant experience of and response to using the ECA | 30 days
  Open- and close-ended questions regarding participant experience of the ECA and response to its use

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study, IPD available by direct request to the PI.

REFERENCES:
- [Result] Magnani JW, Schlusser CL, Kimani E, Rollman BL, Paasche-Orlow MK, Bickmore TW. The Atrial Fibrillation Health Literacy Information Technology System: Pilot Assessment. JMIR Cardio. 2017 Jul-Dec;1(2):e7. doi: 10.2196/cardio.8543. Epub 2017 Dec 12. PMID 29473644
- [Result] Guhl E, Althouse AD, Pusateri AM, Kimani E, Paasche-Orlow MK, Bickmore TW, Magnani JW. The Atrial Fibrillation Health Literacy Information Technology Trial: Pilot Trial of a Mobile Health App for Atrial Fibrillation. JMIR Cardio. 2020 Sep 4;4(1):e17162. doi: 10.2196/17162. PMID 32886070
- [Derived] Guhl EN, Schlusser CL, Henault LE, Bickmore TW, Kimani E, Paasche-Orlow MK, Magnani JW. Rationale and design of the Atrial Fibrillation health Literacy Information Technology Trial: (AF-LITT). Contemp Clin Trials. 2017 Nov;62:153-158. doi: 10.1016/j.cct.2017.09.005. Epub 2017 Sep 18. PMID 28923492